CLINICAL TRIAL: NCT01092234
Title: An Open Randomized Trial of the Effectiveness of an Observational Unit at St. Olavs Hospital
Brief Title: Effectiveness of an Observational Unit at St. Olavs Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2010/105-02; NO883974832 (Other: St.Olavs Hospital)
Record Dates: First submitted 2010-02-23; First posted 2010-03-24 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Emergency Patients
Keywords: Observational units; Length of stay (LOS); Readmission
MeSH Terms: interventions — Organizational Innovation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional ward (Active Comparator)
  Interventions: Other: Traditional ward
- Observational unit (Experimental): Organizational change. Innovative organization of in-hospital care
  Interventions: Other: Organizational change

INTERVENTIONS:
Other: Traditional ward — provision of care in a traditional unit/ward.
  Arms: Traditional ward
Other: Organizational change — Observational unit (new organizational unit) for organizing in-hospital care
  Other Names: Healthcare innovation
  Arms: Observational unit

SUMMARY:
The trial is designed to evaluate the effectiveness of a newly established Observational unit at St. Olavs Hospital in terms of readmission rates, compared to the provision of care in normal/traditional units for defined diagnosis and medical problems.

DETAILED DESCRIPTION:
Observational units are thought to be more efficient than traditional ward units, but the evidence is scarce. The trial will in a randomized fashion evaluate the study hypothesis at an organizational level and not confined to specific diagnosis. The hypothesis to be tested is to confirm or reject the equal effectiveness of an Observational unit compared to a traditional ward for organizing in-hospital care.There are established eligibility and exclusion criteria based on clinical experience. Endpoint is length of stay and readmission within 30 days. In addition the study will give information on the use of diagnostic and treatment resources used and collect some basic demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Emergency admitted patients only
* All patients on the list (appendix 1) with a tentative length of stay < 24 hours
* Predicted stay of less than 24 hours
* Willingness and able to sign a informed consent

Exclusion Criteria:

* Emergency admitted patients with life threatening illnesses
* Patients with a tentative length of stay > 24 hours based on the summary of medical and logistical considerations e.g. need of major - surgery, infections with prolonged infusions of antibiotics.
* Unwillingness to sign a informed consent
* By discretion of the physician/surgeon
* Readmission of any reason in the study period (within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS) | 1 year
  Length of hospital stay in hours

SECONDARY OUTCOMES:
Readmission within 30 days | 30 days
  Readmission to hospital for any reason within 30 calender days

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rødevand, MD, Principal Investigator — St. Olavs Hospital; Siv Mørkved, Professor, Study Chair — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No